CLINICAL TRIAL: NCT00780299
Title: Hemodynamic Efficiency of an Hemodialysis Treatment With High Permeability (HDHP) During the Early Period of Post-resuscitation Shock
Brief Title: Hemodynamic Efficiency of an Hemodialysis Treatment With High Permeability in Post-resuscitation Shock
Acronym: Hyperdia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Gambro Industries, MEYZIEU, France (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071005
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Arrest; Sudden Cardiac Death; Shock
Keywords: Plasma epuration; Hemofiltration; Cardiac arrest; Shock; Inflammatory mediators
MeSH Terms: conditions — Heart Arrest; Death, Sudden, Cardiac; Shock | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): control
  Interventions: Procedure: CVVH
- 1 (Experimental): HDHP
  Interventions: Device: hemodialysis with high permeability (HDHP)

INTERVENTIONS:
Device: hemodialysis with high permeability (HDHP) — HDHP (hemodialysis with high permeability) is a specific plasma epuration of inflammatory mediators
  Arms: 1
Procedure: CVVH — hemofiltration intermittent dialysis
  Arms: 2

SUMMARY:
Rationale: Despite spontaneous cardiac activity recovery, a shock occurs in more than half of patients after resuscitation for cardiac arrest. This acute circulatory insufficiency presents similar characteristics with septic shock and is responsible of most early deaths. Most frequently, usual treatments are unable to control this shock and to avoid the appearance of multiple organ failure.

Aim of the study: In addition to conventional therapeutics, an early plasma epuration of inflammatory mediators (HDHP) could be able to improve hemodynamic parameters and to reduce the shock duration. This improvement could have an impact on multiple organ dysfunctions and also on early mortality.

DETAILED DESCRIPTION:
HDHP (plasma epuration of inflammatory mediators) will be used in addition to the current clinical practice. The experimental arm will be treated by HDHP device.

The high permeability membrane SepteX is a membrane polyarylethersulfone sold by Gambro that allows the purification of molecules of average size to near 50 kd molecular weight.

We can thus purify molecules larger molecular weight than hemofiltration can with the usual membranes (30 kd). Furthermore, this increase in permeability allows a significant treatment medium-sized molecules in diffusion (hemodialysis), that the usual membranes do not allow. Finally, it is possible to purify certain molecules that hemofiltration including high volume does not allow (TNFalpha for example).

Use of this membrane requires the use of specific set dedicated machine Prismaflex itself with a specific software (Exceed) to ensure the control and security of processing.

2 sessions of HDHP will be performed in the first 48 hours following ICU admission (with inclusion in the first 8 hours).

ELIGIBILITY:
Inclusion criteria

* Comatous patients admitted to the ICU for a sudden cardiac death apparently related to heart disease and requiring catecholamine infusion to treat a shock
* Cardiac arrest in front of witnesses
* Written informed consent obtained from the family or by emergency procedure

Exclusion criteria

* Age under 18 years
* Response to verbal commands (Glasgow score >7)
* Terminal illness present before the cardiac arrest
* Acquired or innate immune deficit
* Anticoagulation not recommended or high hemorrhagic risk
* pregnancy
* weight > 100 kg
* without social security
* another clinical trial ongoing
* cardiac arrest from non cardiac etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-11-02 (Actual); Primary Completion 2016-01-02 (Actual); Study Completion 2016-01-02 (Actual)

PRIMARY OUTCOMES:
The main endpoint will be the duration of the shock expressed by the length of catecholamine infusion | 28 days

SECONDARY OUTCOMES:
Changes in organ dysfunction score (SOFA, LOD) during the first 7 days Mortality at day 7 and day 28 Incidence of side effects and complications due to HDHP Impact of HDHP on inflammatory parameters. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Alain Cariou, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Medical intensive care unit of Cochin-St Vincent de Paul university Hospital, Paris, France

REFERENCES:
- [Background] Geri G, Grimaldi D, Seguin T, Lamhaut L, Marin N, Chiche JD, Pene F, Bougle A, Daviaud F, Morichau-Beauchant T, Arnaout M, Champigneulle B, Zafrani L, Bourcier S, Nguyen YL, Charpentier J, Mira JP, Coste J, Vinsonneau C, Cariou A. Hemodynamic efficiency of hemodialysis treatment with high cut-off membrane during the early period of post-resuscitation shock: The HYPERDIA trial. Resuscitation. 2019 Jul;140:170-177. doi: 10.1016/j.resuscitation.2019.03.045. Epub 2019 Apr 8. PMID 30974188